CLINICAL TRIAL: NCT07262931
Title: Effect Of Sensory Motor Training Versus Resistance Training On Improving Pain, Balance And Functional Activities Among Individuals With Knee Osteoarthritis
Brief Title: Effect Of Sensory Motor Training Versus Resistance Training Among Individuals With Knee Osteoarthritis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21657
Record Dates: First submitted 2025-11-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthristis
Keywords: sensory motor training; resistance training; knee osteoarthritis; pain; balance; functional activities
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor remained blinded throughout the study, conducting assessments without knowledge of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Motor Group (Experimental): Participants in the sensory-motor training group received 8-week program of exercise 2 times a week. It starts with a warm-up on stationary bicycle for 10 minutes, stretching exercises.
  Interventions: Other: Sensory motor training
- Resistance training group (Active Comparator): The individuals allocated to the resistance training received a same 8-weeks exercise program twice a week. Exercise began with the same warm-up on stationary bicycle for 10 minutes then traction was applied, Isometric hip flexion and leg extension, stretching exercises for lower limb, Quadriceps and hamstring strengthening using ankle weights were used with frequency twice a week. 3 sets of 10 repetitions at 30 to 40% of 1RM and low to moderate intensity loads were applied for 15 minutes bilaterally.
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Sensory motor training — 7.8. Interventions i FITT Principle: F: 2 times a week I: maximum to minimum T: Group 1 SMT, Group 2 RT T: 40-50 min Individuals were assigned 1:1 to either sensory motor training or resistance training.
  ii Groups with sufficient details
  1 Experimental: Group1: Participants in the sensory-motor training group received 8-week program of exercise 2 times a week. It starts with a warm-up on stationary bicycle for 10 minutes, stretching exercises. In this group the main focus was on agility exercises that includes a balance board, walking on different directions, crossing steps while walking backward and forward and walking on different surfaces. The duration for these exercises was 40-50 minutes per session.
  Arms: Sensory Motor Group
Other: Resistance Training — The individuals allocated to the resistance training received a same 8-weeks exercise program twice a week. Exercise began with the same warm-up on stationary bicycle for 10 minutes then traction was applied, Isometric hip flexion and leg extension, stretching exercises for lower limb, Quadriceps and hamstring strengthening using ankle weights were used with frequency twice a week. 3 sets of 10 repetitions at 30 to 40% of 1RM and low to moderate intensity loads were applied for 15 minutes bilaterally.
  Arms: Resistance training group

SUMMARY:
This study aims to address this gap by comparing the effects of sensory-motor training versus resistance training on pain, balance and functional activities, specifically in patients with early-stage knee osteoarthritis. In Pakistan, Knee Osteoarthritis is a common condition that significantly impacts many individuals' quality of life. While research exists on various exercise interventions for knee osteoarthritis, there is limited focus on patients with Grade 1 and 2 osteoarthritis. Understanding the most effective training method for this group will provide valuable insights for developing targeted rehabilitation programs, ultimately improving patient outcomes and quality of life.

DETAILED DESCRIPTION:
Osteoarthritis of the knee is a degenerative condition that gradually affects the synovial joints. Following the stress, joint become damaged and unable to repair and is triggered by asymmetry in synovial tissues of joint such as articular cartilage, ligaments, subchondral bone, periarticular musculature, menisci, synovia or peripheral nerves. This structural harm leads to the breakdown of subchondral bone and cartilage, resulting in symptoms like stiffness, pain, and limited range of motion. It is just like a plane surface of road becoming uneven and pitted. Osteoarthritis of knee joint debilitates the individuals and they totally rely on others.

Interventions for treating knee osteoarthritis include pharmacological and therapeutic technique. Present clinical recommendations in grade 1 and 2 favor conservative management, like physical therapy, use of assistive devices and weight management due to their simplicity, minimal side effects, and more economical. Due to extensive evidence showing the positive impact of physical activity on individuals with osteoarthritis, exercise is frequently recommended as a key element in the rehabilitation journey.

In various physical workout plans, muscle strengthening holds significance due to the connection between pain, muscle weakness, and limited function. Yet, standard strengthening routines might not suffice for individuals having functional joint instability. A research study on this specific group of patients explored treatments targeting symptoms directly, aiming to enhance the efficiency of the rehabilitation regimen. Recently awareness has been given by focusing on sensory inputs such as balance and proprioception exercises. It may allow individual to adapt motor skills for dealing with disability on knee. Sensorimotor training is an effective treatment to restore motor programs in patients among different musculoskeletal disorders and chronic musculoskeletal pain. It adopts a phase-oriented treatment approach and consists of regulation of arousal, emotion and behavior.

The goal of sensorimotor therapy training in knee osteoarthritis is to gain functional activities, relieve pain. As osteoarthritis advances, sensory-motor abilities like neuromuscular control, static and dynamic balance, and proprioception decrease due to reduced daily physical activities and heightened pain perception. Therefore, incorporating agility, coordination, and balance exercises such as cross steps while walking backward, walking on unsymmetrical surfaces and verbal commands by therapist can be beneficial by challenging individuals with disruptive loads. This exposure helps the neuromuscular system adapt to situations that may trigger knee instability during daily activities. Resistance training refers to a workout method where muscles are engaged against a resistance or weight. This training approach aids in strength enhancement, muscle building, and endurance improvement. It encompasses utilizing weights, resistance bands, or engaging in bodyweight exercises. The benefits of resistance training include overall fitness enhancement, bone density improvement, metabolism boost, and better physical performance. Proper execution of resistance training is crucial to prevent injuries and optimize workout effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Both males and females are included.
* Age group include 40-60 years.
* Not done any exercise for at least 3 months
* Tibiofemoral osteoarthritis
* Grade I and II osteoarthritis

Exclusion Criteria:

* • Cardiorespiratory diseases.

  * Uncontrolled diabetes and Hypertension.
  * Using ambulatory devices.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS - Pain Outcome) | 8 weeks
  The Visual Analogue Scale is a simple, reliable tool used to quantify pain intensity on a 10 cm line ranging from "no pain" to "worst possible pain." Participants marked their pain level experienced in both knees over the past 24 hours.
  It allows sensitive detection of even small changes in perceived pain.
WOMAC Scale (Functional Activities Outcome) | 8 weeks
  The WOMAC Index is a validated questionnaire designed to evaluate pain, stiffness, and physical function specifically in individuals with knee or hip osteoarthritis.
  It assesses daily functional limitations such as walking, stair climbing, and standing.
  Higher scores indicate greater impairment, making it useful for monitoring treatment-related improvements.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Test - Balance Outcome | 8 Weeks
  The Timed Up and Go test measures functional mobility, dynamic balance, and fall risk by timing how long a person takes to stand up from a chair, walk 3 meters, turn, return, and sit down.
  It is quick, practical, and widely used in clinical settings. Longer completion times indicate poorer balance and mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore UBAS, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriacchi TP, Favre J, Erhart-Hledik JC, Chu CR. A systems view of risk factors for knee osteoarthritis reveals insights into the pathogenesis of the disease. Ann Biomed Eng. 2015 Feb;43(2):376-87. doi: 10.1007/s10439-014-1117-2. Epub 2014 Sep 16. PMID 25224078
- [Background] Gomiero AB, Kayo A, Abraao M, Peccin MS, Grande AJ, Trevisani VF. Sensory-motor training versus resistance training among patients with knee osteoarthritis: randomized single-blind controlled trial. Sao Paulo Med J. 2018 Jan-Feb;136(1):44-50. doi: 10.1590/1516-3180.2017.0174100917. Epub 2017 Dec 7. PMID 29236934